CLINICAL TRIAL: NCT04528654
Title: Feasibility of a Web-based Platform to Conduct RCTs of mHealth Apps for CV Risk Factors: Trial My App Hypertension RCT
Brief Title: A Web-based Platform to Conduct Trials of mHealth Apps for Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges in recruitment
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8039
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Risk Factor; Hypertension
Keywords: mobile health; mhealth
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using a web-based blocked randomization list and a 1:1 allocation ratio to one of two possible groups, an intervention group or an educational control group.
Who Masked: Participant
Masking Description: Participants are unblinded. Participants will know if they were assigned to the intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention App Group (Experimental): The intervention group will be instructed to download the chosen hypertension mobile health app (Sphygmo BP) via a link provided on the platform. The hypertension app has blood pressure tracking and monitoring features and they are instructed to use the app. They will also receive a link to the Heart and Stroke foundation website which includes information on hypertension management and measuring blood pressure.
  Interventions: Other: Mobile Health Application
- Educational Control Group (No Intervention): The control will comprise usual care including any anti-hypertensive medication and lifestyle changes, and the link to the Heart and Stroke Foundation website which includes information on hypertension management and measuring blood pressure.

INTERVENTIONS:
Other: Mobile Health Application — The participants will be given instructions to use their smartphone or tablet to download the hypertension tracking app. They will follow the instructions provided within the app and use it to track their blood pressure over the next six months.
  Other Names: Sphygmo BP
  Arms: Intervention App Group

SUMMARY:
Self-management of cardiovascular (CV) risk factors is a recommended form of secondary disease prevention. There are thousands of consumer-facing mobile health (mHealth) applications (apps) intended for tracking, monitoring, and communicating risk factors and health conditions such as hypertension. mHealth apps may be beneficial in improving health status and reducing risk factors. However, the majority of mHealth apps available for consumers have not been scientifically and rigorously evaluated in clinical trials, and due to the fast pace of technological development, those previously evaluated are often outdated by the time trial results are available. Given the rapid pace of change in this field, it is not feasible to rigorously evaluate mHealth apps with current methodologies. McMaster University Health Information Research Unit has developed an innovative research approach using a web-based platform, called Trial My App (TMA), designed to perform efficient, cheap, but high-quality testing of apps relevant to patients with CV risk factors. The overall aim of this pilot study is to test the feasibility of using the web research platform to conduct efficient and rigorous online randomized controlled trials (RCTs) of mHealth apps relevant to patients with CV risk factors. Screening, consent, randomization, and collection of outcomes are completed online using the TMA platform. Recruitment, retention, and completion statistics will be collected in this pilot trial evaluating an mHealth app that targets hypertension. The investigators will partner with clinics in the community to recruit patients to the platform. Study findings will determine if it is feasible to use the relatively simple TMA web-based approach to evaluating the clinical efficacy of mHealth apps for patients with CV risk factors.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of the newly developed Trial My App platform to conduct an efficient RCT of an mHealth app that targets hypertension, a CV risk factor, without the need for in-person visits. Trial stages, including screening, consent, randomization, and collection of patient-important outcomes, will be performed virtually using the TMA platform. A combination of passive and active recruitment will begin in fall 2020 after ethics approval. A variety of recruitment materials will be distributed by a research assistant to partner newsletters, websites, community practices and primary care or speciality clinic waiting rooms. These materials include videos, paper and online posters/postcards, emails, as well as posts advertising on social media. Social media recruitment will consist of general posts and targeted ads. The primary goal at this stage is to determine whether TMA, the innovative, efficient, web-based methodology, can be used to conduct RCTs evaluating mHealth interventions. The primary feasibility outcome is study completion. Other feasibility outcomes are recruitment rate, eligibility rates, consent rates, retention rates, intervention adherence, and appropriateness of data collection processes. Descriptive analysis will be performed on the dataset using appropriate statistical methods. The secondary objective is to test the clinical efficacy of the chosen mHealth app in reducing BP in patients with sub-optimally controlled hypertension when compared with an educational control group. Efficacy outcomes include clinical assessment changes, self-management adherence, and patient-reported outcomes. This is a pilot, non-blinded, feasibility RCT, comparing use of a hypertension tracking app versus an education control in participants with hypertension that is sub optimally controlled. The investigators will later include a sub-study to validate the blood pressure data inputted into the online platform through in-person blood pressure measurements. Participants will be asked to register on the TMA site and will complete user profile and screening questionnaires and consent for participation in the pilot trial. The participants that meet inclusion criteria will be asked to electronically consent to take part in the pilot trial, and input clinical and patient-important data at 0, 1, 3, and 6 months into the web application.

ELIGIBILITY:
Inclusion Criteria

* age over 18
* diagnosis of hypertension
* interested in using an app for hypertension management
* access to a smartphone with internet connection
* access to a blood pressure monitoring device (in home or community setting, e.g., pharmacy)

Exclusion Criteria:

* participant-reported BP within target within the 2 weeks prior to enrolment. Target range for patients with diabetes is systolic BP <130 mm Hg and diastolic BP < 80 mm Hg; for those without diabetes, target range is systolic BP <140 mm Hg and diastolic BP < 90 mm Hg according to Hypertension Canada guidelines
* emergent hypertensive concerns with systolic BP ≥180 mmHg or diastolic BP ≥120 within the 2 weeks prior to enrolment
* current use of a mobile app for hypertension management
* pregnancy
* not living in Canada
* unwillingness or inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Participation completion | 6-months
  Proportion of registered participants who successfully complete the 6-month questionnaire

SECONDARY OUTCOMES:
Change from baseline blood pressure at 6 months | Baseline, 6-months
  Statistically significant difference in mean change in systolic BP measurements [defined as P<0.05 using a Pearson test] compared to standard ranges from baseline to six months between groups.
Change from baseline self-management adherence at 6 months | Baseline, 6-months
  Differences in mean change to adherence to hypertension self-care behaviors. This will be scored using the H-SCALE.
Change from baseline healthcare self-efficacy at 6 months | Baseline, 6-months
  Differences in mean change to healthcare self-efficacy. This will be scored using the frequency distribution and mean of the Health Confidence Score, a 4-item Likert scale.
Change from baseline patient-reported outcomes at 6 months | Baseline, 6-months
  Descriptive analysis of patient-oriented experiences between groups measured in a 5-point Likert scale questionnaire developed from advisory board themes at 95% confidence interval (CI)
Eligibility rate | Baseline
  The number of patients meeting eligibility criteria in baseline and screening questionnaires.
Consent rate | Baseline
  The proportion of eligible participants consenting to participating in the trial with an electronically signed consent form.
Retention rate | 6-months
  The proportion of withdrawals and drop-outs post-recruitment.
Outcome acceptability | 6-months
  Proportion of questionnaires completed and submitted
Appropriateness of data collection processes | 6-months
  Completeness and accuracy of data in each questionnaire
Recruitment rate | Baseline
  The number of patients successfully recruited to the platform
Change from baseline intervention acceptability at 6 months | Baseline, 6-months
  Frequency of app usage between control and intervention groups based on answers to questionnaires
Concordance of self-reported blood pressure | 6-months
  Concordance between self-reported blood pressure readings and in-person collected data

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Lokker, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Lokker C, Jezrawi R, Gabizon I, Varughese J, Brown M, Trottier D, Alvarez E, Schwalm JD, McGillion M, Ma J, Bhagirath V. Feasibility of a Web-Based Platform (Trial My App) to Efficiently Conduct Randomized Controlled Trials of mHealth Apps For Patients With Cardiovascular Risk Factors: Protocol For Evaluating an mHealth App for Hypertension. JMIR Res Protoc. 2021 Feb 1;10(2):e26155. doi: 10.2196/26155. PMID 33522978